CLINICAL TRIAL: NCT02616718
Title: Incisional Hernia Progression Over Time
Acronym: INPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Kristian Kiim Jensen, MD, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-15008340
Record Dates: First submitted 2015-11-21; First posted 2015-11-30 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Hernia, Ventral
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ventral incisional hernia (Experimental): Repeated computed tomography scan of abdomen
  Interventions: Radiation: Repeated computed tomography scan of abdomen

INTERVENTIONS:
Radiation: Repeated computed tomography scan of abdomen — Repeated computed tomography scan of abdomen within two weeks prior to surgery or 28-32 weeks after initial scan

SUMMARY:
This is a prospective multicenter study of patients diagnosed with a medium to giant incisional hernia (transverse defect >7 cm). Patients referred to the surgical outpatient clinic are invited to participate in the study. As a standard, all patients who are examined for incisional hernia undergo CT scan according to a hernia protocol, before planning of surgical repair (baseline scan). After this CT scan, patients are seen in the out-patient clinic once again and either treated conservatively without surgery, or scheduled for elective surgical repair of the hernia.

If surgery is planned, the patients participating in the study undergo an additional CT scan in hernia protocol, within two weeks prior to surgery (follow-up scan).

If a conservative non-surgical approach is chosen, patients can still participate in the study and will undergo an additional CT scan after 28-32 weeks.

DETAILED DESCRIPTION:
This is a prospective multicenter study of patients diagnosed with a medium to giant incisional hernia (transverse defect >7 cm). Patients referred to the surgical outpatient clinic are invited to participate in the study. As a standard, all patients who are examined for incisional hernia undergo CT scan according to a hernia protocol, before planning of surgical repair (baseline scan). After this CT scan, patients are seen in the out-patient clinic once again and either treated conservatively without surgery, or scheduled for elective surgical repair of the hernia.

If surgery is planned, the patients participating in the study undergo an additional CT scan in hernia protocol, within two weeks prior to surgery (follow-up scan). In case no baseline scan in hernia protocol exists, patients will undergo this scan immediately after inclusion in the study. Furthermore, patients will be asked to fill out a questionnaire on physical activity (IPAQ) and hernia-related quality of life (HerQLes) at the time of the baseline and follow-up scans. IPAQ is a well-validated questionnaire, which assesses patients' physical activity within the last 7 days. The outcome is metabolic minutes per week, a numerical value which places the responder in one of three categories: Low, moderate or high physical activity. HerQLes is a validated questionnaire assessing the hernia-related quality of life. This questionnaire has been translated into Danish using a standardized protocol. The outcome is a numerical score of 0-100, with 100 being the highest hernia-related quality of life. Currently, the time from planning of hernia repair to surgery is approximately 30 weeks. Thus, the mean time between the two CT scans should be around 28-32 weeks.

If a conservative non-surgical approach is chosen, patients can still participate in the study and will undergo an additional CT scan after 28-32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Suspected incisional hernia with a horizontal fascial defect > 7 cm

Exclusion Criteria:

* Inability to read or speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Fascial defect area | 28-32 weeks
  Change fascial defect area from initial CT scan to follow-up CT scan

SECONDARY OUTCOMES:
Hernia-related quality of life | 28-32 weeks
  Change in Hernia-related quality of life
Physical activity | 28-32 weeks
  Change in physical activity, measured by International Physical Activity Questionnaire
Hernia sac volume | 28-32 weeks
  Change in hernia sac volume measured on repeated CT scans

CONTACTS AND LOCATIONS:
Overall Officials: Kristian K Jensen, MD, Principal Investigator — Bispebjerg Hospital, University of Copenhagen
Locations (1):
- Digestive Disease Center, Bispebjerg Hospital, Copenhagen NV, Copenhagen, Denmark